CLINICAL TRIAL: NCT00441025
Title: A Phase II Study of Alemtuzumab in Combination With CHOP as First-Line Treatment in Peripheral T-Cell Lymphoma
Brief Title: The Effectiveness of Alemtuzumab Combination With CHOP to Treat Patients Newly Diagnosed With PTCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: a lack of a potential patient.
Sponsor: Mahidol University (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH 011002
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2007-02

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: MabCampath + CHOP in PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Alemtuzumab

ARMS (1):
- 1 (Active Comparator): 1 Alemtuzumab
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab

SUMMARY:
The purpose of this study is to determine whether the treatment of Alemtuzumab in combination with CHOP(cyclophosphamide,doxorubicin,vincristine and prednisolone) are effective as first line treatment in patients with peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) are more common in Asia than in Europe and United States (17-40% vs. 5-10%). Most studies reported a poorer prognosis for PTCL compared to B-cell non-Hodgkin's lymphomas (NHL).

CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) is currently regarded as a standard chemotherapy regimen for patients with newly diagnosed NHL.

Alemtuzumab (Campath-1H) is a humanized monoclonal antibody that targets CD52, a cell surface protein present at high density on most normal and malignant B and T lymphocytes.Malignant T cells express particularly high numbers of CD52 cell surface markers (approximately 500,000 molecules/lymphocytes),T-cell malignancies may thus be particularly responsive to alemtuzumab.

As the response rate tend to be higher in patients newly diagnosed with PTCL, this study evaluates the efficacy of alemtuzumab in combination with CHOP administered as up-front therapy in patients newly diagnosed with PTCL in terms of response rate and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following histologic types according to the WHO classification:

  * Angioimmunoblastic T-cell lymphoma
  * Extranodal NK/T-cell lymphoma,nasal type
  * Enteropathy-type T-cell lymphoma
  * Hepatosplenic gamma-delta T-cell lymphoma
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Anaplastic large-cell lymphoma,T/null cell,primary systemic type
  * Peripheral T-cell lymphoma,not otherwise characterized
* Newly diagnosed,age 15-65 years.
* Complete work up for baseline evaluation and measurement (Appendix B)
* Patient's free written inform consent.

Exclusion Criteria:

* Patients with a known hypersensitivity to murine proteins or to any component of alemtuzumab.
* Patients who have received prior antilymphoma treatment with chemotherapy or radiotherapy
* Patients with poor performance status (PS;ECOG criteria of 3-4)(Appendix C).
* Serologic evidence of HCV and HCV RNA of chronic hepatitis.
* Serologic evidence of HBV and HBV RNA of chronic hepatitis.
* Patients with history of impaired cardiac status or myocardial infarction.
* Patients with serum creatinine >= 1.8 mg/dl,bilirubin >= 1.5 times upper limit of normal range,SGOT or SGPT >= 3 times upper limit of normal range, unless due to tumor involvement.
* Patients with active uncontrolled infection,active non-malignant gastric or duodenal ulcer, uncontrolled diabetes mellitus or other severe medical conditions which would preclude aggressive cytotoxic chemotherapy.
* Active secondary malignancy.
* Pregnant or lactating women.
* Serious medical or psychiatric illness which prevent informed consent.
* Patients who are likely to lost to follow up (eg, unwilling or difficult to return,cannot be contacted).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-09; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of alemtuzumab given in combination with CHOP in terms of the rates of objective response rate (ORR:complete remission[CR] and
partial remission[PR]),progressive disease-free(PFS) and overall survivals(OS)
in patients newly diagnosed with PTCL.

SECONDARY OUTCOMES:
To determine the safety profiles of alemtuzumab given in combination with CHOP

CONTACTS AND LOCATIONS:
Overall Officials: Surapol Issaragrisil, M.D.,Prof., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand